CLINICAL TRIAL: NCT06736899
Title: Randomized Trial of Orbital Atherectomy Versus Standard Strategy in Calcified Bifurcation Lesions
Brief Title: Trial of Orbital Atherectomy Versus Standard Strategy in Calcified Bifurcation Lesions
Acronym: OraBil
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación EPIC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EPIC44-OraBil
Record Dates: First submitted 2024-12-11; First posted 2024-12-17 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Coronary Artery Disease; Coronary Disease
Keywords: Orbital Atherectomy (OA); Percutaneous Coronary Intervention; Bifurcation; Side Branch Treatment: Mid-term results
MeSH Terms: conditions — Coronary Artery Disease; Coronary Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Balloon Angioplasty (BA) (Active Comparator)
  Interventions: Device: Balloon System Treatment
- Orbital Atherectomy (OA) (Active Comparator)
  Interventions: Device: Orbital Atherectomy System Treatment

INTERVENTIONS:
Device: Orbital Atherectomy System Treatment — Percutaneous coronary intervention of a calcified bifurcation coronary lesion with balloon angioplasty followed by drug eluting stent. Selection of balloon type is at operator´s discretion. Baseline and post dilation OCT will be performed.
  Arms: Orbital Atherectomy (OA)
Device: Balloon System Treatment — Percutaneous coronary intervention of a calcified bifurcation coronary lesion with Orbital Atherectomy followed by drug eluting stent. Baseline and post dilation OCT will be performed.
  Arms: Balloon Angioplasty (BA)

SUMMARY:
Clinical research with medical devices indicated in accordance with the CE marking, led by researchers, multicenter, open, prospective, randomized and controlled. Patients are randomized to treatment with a conventional balloon and then a coronary stent or to initial plaque modification with Orbital Atherectomy (OA) and then a coronary stent. To evaluate the efficacy and safety of OA in the adequate treatment with coronary stent of the calcified bifurcation lesion using angiography and optical coherence tomography (OCT).

DETAILED DESCRIPTION:
The risk profile of patients and their comorbidities have worsened and the observed lesions undergoing treatment are increasingly complex. This has promoted the development of new technologies for plaque modification, especially in the context of calcified lesions. These predispose to suboptimal results of the intervention due to an increased risk of malapposition and underexpansion of the stents, the main variables for restenosis and/or thrombosis of the stents. Thus, compared with non-calcified lesions, the increased amount of calcium in the coronary artery leads to a higher incidence of major adverse cardiac events (MACE).

Coronary bifurcation stenting remains complex and is associated with a high risk of stent thrombosis and restenosis even with contemporary techniques, and suboptimal outcomes are frequently observed due to side branch (SL) involvement that increases cardiovascular events.

Our hypothesis is that the use of orbital atherectomy (OA) for coronary revascularization in the presence of calcified bifurcation lesions is feasible and safe compared to the more common technique, favoring the subsequent performance of provisional stenting (PS).

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age and
* Patients with moderately or severely calcified bifurcation lesions (lateral vessel ≥ 2mm), candidates for PCI with coronary stent implantation, in whom there is the possibility of adequate clinical follow-up at 1 year and
* Patients agree to participate in the study, by signing the Informed Consent.

Exclusion Criteria:

* Patients with revascularization of the artery to be treated within 9 months prior to the index procedure.
* Patients with contraindication for the use of Orbital Atherectomy:

  * Patients in cardiogenic shock.
  * Patients with Thrombotic lesions.
  * Patients with Vascular graft disease.
  * Patients with remain vessel disease.
  * Patients with severe left ventricular dysfunction.
  * Patients allergic to the components of the washing serum (glide).
* Patients with life expectancy less than one year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-10-23 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
EFFICACY: Angiographic criteria success | At the end of PCI (Percutaneous Coronary Intervention)
  Percentage of Main vessel and side branch (≥2 mm) patency (final stenosis <20%) without the presence of: residual lesion >70% and TIMI flow < 3 and residual ≥ type C disection
EFFICACY: OCT criteria: Stent expansion | At the end of PCI
  Percentage of MLA / mean reference luminal area (mean proximal and distal reference luminal)

SECONDARY OUTCOMES:
SAFETY:Major adverse cardiac events (MACE) | 12 months
  Rate of cardiac death, myocardial infarction (MI), target lesion revascularization (TLR), and non-target lesion target vessel revascularization (TVR non-TLR), thrombosis and stroke
SAFETY:Major adverse cardiac events (MACE) | 6 months
  Rate of cardiac death, myocardial infarction (MI), target lesion revascularization (TLR), and non-target lesion target vessel revascularization (TVR non-TLR), thrombosis and stroke
SAFETY:Major adverse cardiac events (MACE) | 30 days
  Rate of cardiac death, myocardial infarction (MI), target lesion revascularization (TLR), and non-target lesion target vessel revascularization (TVR non-TLR), thrombosis and stroke
SAFETY:Major adverse cardiac events (MACE) | At the end of PCI
  Rate of cardiac death, myocardial infarction (MI), target lesion revascularization (TLR), and non-target lesion target vessel revascularization (TVR non-TLR), thrombosis and stroke
EFFICACY: Other variables related to stent expansion. Minimal Lumen Area (MLA) in mm2 | At the end of PCI
  Cut-off point >5 mm2
EFFICACY: Other variables related to stent expansion. Minimal Lumen Area (MLA) | At the end of PCI
  Percentage of Cut-off point >90 mm2
EFFICACY: Other variables related to stent expansion. Mean stent expansion | At the end of PCI
  Percentage of mean stent area (sum of stent area/analyzed stent length)/mean reference lumen area (cut-off point>80%)
EFFICACY: Other variables related to stent expansion. Stent expansion using linear model | At the end of PCI
  Percentage of stent volume/adaptative reference lumen volume. (cut-off point>65%)

CONTACTS AND LOCATIONS:
Locations (3):
- Spain (3):
  - H. G.U. de ALICANTE DR. BALMIS, Alicante
  - Hospital Universitario Lucus Augusti, Lugo
  - Hospital Universitario La Luz, Madrid

REFERENCES:
- [Background] Parikh K, Chandra P, Choksi N, Khanna P, Chambers J. Safety and feasibility of orbital atherectomy for the treatment of calcified coronary lesions: the ORBIT I trial. Catheter Cardiovasc Interv. 2013 Jun 1;81(7):1134-9. doi: 10.1002/ccd.24700. Epub 2013 Mar 5. PMID 23460596
- [Background] Burzotta F, Louvard Y, Lassen JF, Lefevre T, Finet G, Collet C, Legutko J, Lesiak M, Hikichi Y, Albiero R, Pan M, Chatzizisis YS, Hildick-Smith D, Ferenc M, Johnson TW, Chieffo A, Darremont O, Banning A, Serruys PW, Stankovic G. Percutaneous coronary intervention for bifurcation coronary lesions using optimised angiographic guidance: the 18th consensus document from the European Bifurcation Club. EuroIntervention. 2024 Aug 5;20(15):e915-e926. doi: 10.4244/EIJ-D-24-00160. PMID 38752714
- [Background] den Dekker WK, Siskos AA, Wilschut JM, Nuis RJ, Scarparo P, Neleman T, Masdjedi K, Ligthart JMR, Diletti R, Daemen J, Van Mieghem NM. Initial experience with orbital atherectomy in a tertiary centre in the Netherlands. Neth Heart J. 2023 May;31(5):196-201. doi: 10.1007/s12471-022-01742-3. Epub 2022 Dec 12. PMID 36507948
- [Background] Donatelle M, Agasthi P, Parise H, Igyarto Z, Martinsen BJ, Leon MB, Beohar N. Coronary Orbital Atherectomy in Patients With Severe Aortic Stenosis. J Invasive Cardiol. 2022 Oct;34(10):E696-E700. doi: 10.25270/jic/22.00066. PMID 36200995
- [Background] Jurado-Román A, Gómez-Menchero A, Gonzalo N, et al. Plaque modification techniques to treat calcified coronary lesions. Position paper from the ACI-SEC. REC Interv Cardiol Engl Ed. Published online February 7, 2023:9672. doi:10.24875/RECICE.M22000345